CLINICAL TRIAL: NCT06499766
Title: Methodological Study of the Effect of a Lotion Containing Nature Based Microbial Extract on Atopic Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uute Scientific Oy (Industry)
Collaborators: Tampere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Uuteatopia1
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Atopic Dermatitis
Keywords: Biodiversity intervention; Allergy; Microbes
MeSH Terms: conditions — Dermatitis, Atopic; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Lotions looks the same. Participants, investigators or outcome assessors don't know which lotion (placebo or active ingredient) is used in which arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature-based exposure by biodiversity component in lotion. (Active Comparator): Biodiversity component is highly diverse microbial extract mimicking Finnish forest soil biodiversity. Component is added to the common moisturizer on the Finnish market.
  Interventions: Other: Biodiversity intervention by inactivated microbial extract
- Placebo by coloring component in lotion. (Placebo Comparator): Coloring ingredient is safe, biochemically non-active component which purpose is to make the placebo lotion looking same as the biodiversity lotion in other arm. Component is added to the common moisturizer on the Finnish market (same as in the other arm).
  Interventions: Other: Placebo intervention by colored lotion

INTERVENTIONS:
Other: Biodiversity intervention by inactivated microbial extract — Participants use the lotion including microbial extract on one arm twice a day for 28 days. No other lotions or creams are used simultaneously on this area. Atopy medicines are not used during the trial or 14 days before the trial.
  Arms: Nature-based exposure by biodiversity component in lotion.
Other: Placebo intervention by colored lotion — Participants use the lotion including safe, non-active coloring ingredient on one arm twice a day for 28 days. No other lotions or creams are used simultaneously on this area. Atopy medicines are not used during the trial or 14 days before the trial.
  Arms: Placebo by coloring component in lotion.

SUMMARY:
The purpose of the study is to test the selected methods and to explore the effect of nature-based exposure on immunological biomarkers and the condition of atopic skin. Overall purpose is to test the safety and feasibility of a new nature-exposure method on atopic skin: regular use of lotion containing inactivated microbial extract that mimics Finnish forest microbial biodiversity.

DETAILED DESCRIPTION:
According of hygiene and biodiversity hypotheses, regular contact to nature biodiversity is beneficial for human health. Without the contact, there is risk for immune system malfunction and related diseases like atopy, allergies and inflamed bowel diseases. Regular contact to natural biodiversity, including environmental microbes, add immunological tolerance and train immune system to separate dangerous external stimuli from non-dangerous ones.

This study aim at testing if it is safe to use microbial extract in lotion on daily basis on atopic skin. Study participants are adults and they have atopic dermatitis diagnosis. Participants use the lotion with microbial extract on other arm and placebo lotion (same lotion but microbial extract is replaced with safe coloring ingredient) on the other arm two times per day for 28 days. Atopy medicines are not used on the study period and 14 days before the study. Also, other moisturizers than test lotions are not used on test areas during the study.

Study is placebo controlled, randomized and double-blinded.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65
* Legally competence
* Fullfills Hanifin & Rajka criteria for atopic dermatitis
* Commitment to the study

Exclusion Criteria:

* Regular contact to farming environment
* Cancer or on going cancer treatments
* Use of immunosuppressive medicines
* Photo therapy, solarium or vacation abroad during the study
* Too severe eczema (not possible to keep pause from atopy medicines)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Transepidermal water loss (TEWL) | 0, 14 and 28 days
  TEWL measurement from each test area (arms)

SECONDARY OUTCOMES:
Skin erythema index | 0, 14 and 28 days
  Erythema index measurement from each test area (arms)
SCORAD (SCORing Atopic Dermatitis) | 0 and 28 days
  Scoring of atopic dermatitis (whole body) by dermatologist. Scale 0-103.
Local scoring of eczema on arms | 0 and 28 days
  Local scoring of eczema only on arms (each arm separately) by dermatologist. Scale 0-18.
Pro-inflammatory cytokines on skin | 0 and 28 days
  Tape strip samples from both arms and cytokine analysis from the samples.
Self evaluation of eczema symptoms and effect of the lotion | 0, 7, 14, 21 and 28 days
  Filling of self questionnaire every week

CONTACTS AND LOCATIONS:
Locations (1):
- Uute Scientific Oy, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No